CLINICAL TRIAL: NCT00588783
Title: I-beam and Cruciate Tibial Components Used in Total Knee Replacement
Status: Terminated | Type: Observational
Sponsor: Biomet Orthopedics, LLC (Industry)
Collaborators: New Lexington Clinic (Other)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Other Study IDs: 104-U-013
Record Dates: First submitted 2007-12-21; First posted 2008-01-09 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Degenerative Arthritis; Osteoarthritis; Rheumatoid Arthritis; Knee Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
  Interventions: Device: I-beam design
- 2
  Interventions: Device: Cruciate design

INTERVENTIONS:
Device: I-beam design — This group will utilize tibial components with an I-beam design for total knee replacement.
  Groups: 1
Device: Cruciate design — This group will utilize tibial components with cruciate designs for total knee replacement.
  Groups: 2

SUMMARY:
The purpose of this study is to compare the clinical outcomes of using an I-beam or cruciate tibial component in total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful and disabled knee joint resulting from osteoarthritis, rheumatoid arthritis, traumatic arthritis where one or more compartment are involved.
* Patients requiring correction of varus, valgus, or posttraumatic deformity
* Patients requiring correction of revision of unsuccessful osteotomy, arthrodesis, or failure of previous joint replacement procedure.

Exclusion Criteria:

* Patients with infection, sepsis, or osteomyelitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients requiring total knee replacement.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Revision rate | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Biomet Orthopedics, LLC, Warsaw, Indiana, United States